CLINICAL TRIAL: NCT00140595
Title: Randomized Study of ACVBP Plus Rituximab Versus CHOP Plus Rituximab in Patients Aged From 18 to 59 Years With Diffuse Large B-cell Lymphoma and a Age-adjusted IPI of 1.
Brief Title: ACVBP Plus Rituximab Versus CHOP Plus Rituximab in Patients With Diffuse Large B-cell Lymphoma and Age-adjusted IPI of 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Amgen (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNH03-2B
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Diffuse Large-Cell Lymphoma
Keywords: Lymphoma, diffuse large B-cell; rituximab; chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: rituximab
Drug: doxorubicin
Drug: cyclophosphamide

SUMMARY:
This study is a multicentric randomized trial evaluating the efficacy of the combination ACVBP+rituximab compared to the combination of CHOP+rituximab in patients aged from 18 to 59 years with diffuse large B-cell lymphoma and one factor of the age-adjusted international prognostic index (IPI).

DETAILED DESCRIPTION:
This phase III multicentric open label randomized study is based on the results of previous LNH 93-5 and LNH98-5 studies.

The LNH93-5 study has shown that the ACVBP regimen gave a longer EFS (39% vs 29% at 5 years, p=0.005) and a longer overall survival (46% vs 38% at 5 years, p=0.036) than CHOP in patients aged between 61 and 69 with an IPI score ≥1. However ACVBP had a more important toxicity and a higher treatment related mortality (13% vs 7%, p<0.01), specially after 65 years. In younger patients ACVBP is better tolerated.

The addition of Rituximab to standard CHOP (R-CHOP) has been shown in LNH98-5 study to improve complete remission rate (CR), event-free survival (EFS) and overall survival (OS) in elderly patients with B-DLCL. Considering only patients with an aa-IPI score of 1, the 2 year EFS was 75% in the R-CHOP group as compared with 42% in the CHOP group.

This study is designed to test whether addition of rituximab to ACVBP is better than R-CHOP in patients younger than 60. Primary endpoint is event-free survival, we expect a gain in 2 years-EFS of 10% in R-ACVBP group as compared with R-CHOP group.

This study is a multicentric, phase III open-label, randomized trial evaluating the efficacy of ACVBP+rituximab compared to CHOP+rituximab in patients aged from 18 to 59 years with non previously treated diffuse large B-cell lymphoma and one factor of the age-adjusted international prognostic index

ELIGIBILITY:
Inclusion Criteria:

Patient with histologically proven CD20+ diffuse large B-cell lymphoma (WHO classification) Aged from 18 to 59 years. Age-adjusted International Prognostic Index equal to 1 (elevated LDH level OR stage III-IV OR ECOG status 2-3-4).

Patient not previously treated. With a minimum life expectancy of 3 months. Negative HIV, HBV and HCV serologies test 4 weeks (except after vaccination). Having previously signed a written informed consent.

Exclusion Criteria:

Any other histological type of lymphoma. Any history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included.

Central nervous system or meningeal involvement by lymphoma. Contra-indication to any drug contained in the chemotherapy regimens. Any serious active disease (according to the investigator's decision). Poor renal function (creatinin level>150µmol/l), poor hepatic function (total bilirubin level>30mmol/l, transaminases>2.5 maximum normal level) unless these abnormalities are related to the lymphoma.

Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration.

Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.

Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.

Pregnant or lactating women. Adult patient under tutelage.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Estimated)
Dates: Start 2003-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS), events defined as death from any cause, relapse for complete responders (CR) and unconfirmed complete responders (CRu), progression during or after treatment, changes of therapy during allocated treatment.

SECONDARY OUTCOMES:
Response rate at the end of the treatment, progression rate, relapse rate, disease-free survival for complete responders, overall survival, neuromeningeal relapse rate and additional toxicities with ACVBP+rituximab combination

CONTACTS AND LOCATIONS:
Overall Officials: Christian Recher, MD, Principal Investigator — Lymphoma Study Association; Hervé Tilly, MD, Study Chair — Lymphoma Study Association; Corinne Haioun, MD, Study Chair — Lymphoma Study Association
Locations (10):
- Groupe d'étude des lymphomes de l'adulte, Yvoir, Belgium
- France (9):
  - Hôpital Henri Mondor, Créteil
  - Centre Léon Bérard, Lyon
  - Hôpital Saint Louis, Paris
  - Hématologie Adultes - Hôpital Necker, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Hématologie CHU Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Tilly H, Lepage E, Coiffier B, Blanc M, Herbrecht R, Bosly A, Attal M, Fillet G, Guettier C, Molina TJ, Gisselbrecht C, Reyes F; Groupe d'Etude des Lymphomes de l'Adulte. Intensive conventional chemotherapy (ACVBP regimen) compared with standard CHOP for poor-prognosis aggressive non-Hodgkin lymphoma. Blood. 2003 Dec 15;102(13):4284-9. doi: 10.1182/blood-2003-02-0542. Epub 2003 Aug 14. PMID 12920037
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Dumontet C, Mounier N, Munck JN, Bosly A, Morschauser F, Simon D, Marit G, Casasnovas O, Reman O, Molina T, Reyes F, Coiffier B. Factors predictive of early death in patients receiving high-dose CHOP (ACVB regimen) for aggressive non-Hodgkin's lymphoma: a GELA study. Br J Haematol. 2002 Jul;118(1):210-7. doi: 10.1046/j.1365-2141.2002.03565.x. PMID 12100150
- [Derived] Ghesquieres H, Larrabee BR, Haioun C, Link BK, Verney A, Slager SL, Ketterer N, Ansell SM, Delarue R, Maurer MJ, Fitoussi O, Habermann TM, Peyrade F, Dogan A, Molina TJ, Novak AJ, Tilly H, Cerhan JR, Salles G. FCGR3A/2A polymorphisms and diffuse large B-cell lymphoma outcome treated with immunochemotherapy: a meta-analysis on 1134 patients from two prospective cohorts. Hematol Oncol. 2017 Dec;35(4):447-455. doi: 10.1002/hon.2305. Epub 2016 Jun 10. PMID 27282998
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- [Derived] Molina TJ, Canioni D, Copie-Bergman C, Recher C, Briere J, Haioun C, Berger F, Ferme C, Copin MC, Casasnovas O, Thieblemont C, Petrella T, Leroy K, Salles G, Fabiani B, Morschauser F, Mounier N, Coiffier B, Jardin F, Gaulard P, Jais JP, Tilly H. Young patients with non-germinal center B-cell-like diffuse large B-cell lymphoma benefit from intensified chemotherapy with ACVBP plus rituximab compared with CHOP plus rituximab: analysis of data from the Groupe d'Etudes des Lymphomes de l'Adulte/lymphoma study association phase III trial LNH 03-2B. J Clin Oncol. 2014 Dec 10;32(35):3996-4003. doi: 10.1200/JCO.2013.54.9493. Epub 2014 Nov 10. PMID 25385729
- [Derived] Recher C, Coiffier B, Haioun C, Molina TJ, Ferme C, Casasnovas O, Thieblemont C, Bosly A, Laurent G, Morschhauser F, Ghesquieres H, Jardin F, Bologna S, Fruchart C, Corront B, Gabarre J, Bonnet C, Janvier M, Canioni D, Jais JP, Salles G, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte. Intensified chemotherapy with ACVBP plus rituximab versus standard CHOP plus rituximab for the treatment of diffuse large B-cell lymphoma (LNH03-2B): an open-label randomised phase 3 trial. Lancet. 2011 Nov 26;378(9806):1858-67. doi: 10.1016/S0140-6736(11)61040-4. PMID 22118442